CLINICAL TRIAL: NCT02136576
Title: Comparing Three Caries Prevention Products on Dentinal Hypersensitivity - A Pilot Study
Brief Title: Caries Prevention Products & Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Britta Magnuson, Asst. Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11184; New Investigator Grant (Other: TUSDM)
Record Dates: First submitted 2014-05-07; First posted 2014-05-13 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sensodyne (Active Comparator): There are no specific characteristics for inclusion in this group. Enrollment will be determined randomly.
  Interventions: Device: Sensodyne
- Crest Cavity Protection & MI Paste Plus (Active Comparator): There are no specific characteristics for inclusion in this group. Enrollment will be determined randomly.
  Interventions: Device: Crest Cavity Protection & MI Paste Plus
- Clinpro 5000 (Active Comparator): There are no specific characteristics for inclusion in this group. Enrollment will be determined randomly.
  Interventions: Device: Clinpro 5000

INTERVENTIONS:
Device: Sensodyne — Subjects will be instructed to brush with Sensodyne twice daily (2 minutes each time in the morning and the evening) during the duration of the study.
  Arms: Sensodyne
Device: Crest Cavity Protection & MI Paste Plus — Subjects will be instructed to brush twice daily (2 minutes each time in the morning and the evening) using Crest Cavity Protection toothpaste. They will be instructed to apply MI Paste Plus (CPP-ACP with fluoride) twice daily to the study teeth after brushing their teeth. MI Paste Plus will be applied to the study teeth with a finger.
  Arms: Crest Cavity Protection & MI Paste Plus
Device: Clinpro 5000 — Subjects will be instructed to brush with Clinpro 5000 twice daily (2 minutes each time in the morning and the evening) during duration of the study.
  Arms: Clinpro 5000

SUMMARY:
The aim of this pilot research project is to compare the clinical effect on dentinal hypersensitivity of three products: Casein Phosphopeptide-Amorphous Calcium Phosphate (CPP-ACP) paste with fluoride, 5000 Sodium Fluoride (NaF) dentifrice containing Tri-Calcium Phosphate (TCP), and a dentifrice containing Potassium Nitrate.

The hypothesis of this study is that CPP-ACP with fluoride and 5000ppm NaF with TCP will exhibit a greater reduction in dentinal hypersensitivity compared to the control (dentifrice containing Potassium Nitrate).

The results of this pilot study will validate or negate the need for a larger clinical study that may provide generalizable results for using caries-prevention products with the additional benefit of minimizing dentinal hypersensitivity.

DETAILED DESCRIPTION:
Dentinal hypersensitivity commonly occurs in patients with gingival recession, resulting from a reduced periodontium or in patients who have undergone non-surgical and surgical periodontal therapy (Pradeep 2010, Yilmaz 2011). When the gingiva recede, the root surfaces of the teeth are exposed (West 2008). In addition, after a non-surgical or surgical periodontal procedure, the cementum of the root surface is removed as a result of scaling and root planing. This leaves dentin exposed on the root surface with open dentinal tubules. In addition, dentin is less mineralized than enamel and has a greater susceptibility to and a faster progression of root caries and dentinal hypersensitivity (Saunders 2005). Root caries commonly occurs in patients who have undergone periodontal therapy and extensive root caries often results in the extraction of the tooth (Hull 1997).

Dental professionals often make a variety of recommendations to remedy dental hypersensitivity, including the application of fluoride varnishes, anti-hypersensitivity toothpaste, gingival grafting procedures and various restorative procedures, aiming to occlude the dentinal tubules or desensitize the pulpal nerve endings (Brahmbhatt 2012, Orsini 2010).

Since the introduction of Caries Management By Risk Assessment (CAMBRA) in the Journal of the California Dental Association in 2007 (Jenson 2007, Young 2007), the marketplace for anti-caries products has surged. As a result, many approaches to the management of dental caries have been introduced and dental practitioners and sales representatives have promoted several anti-caries products. In addition, the reduction or the abatement of the progression of dental caries (coronal, root and interproximal) as a result of a caries management program has been reported (Featherstone 1992, Ito 2012). Many caries management products have ingredients that include fluoride and calcium phosphate (Amorphous Calcium Phosphate-Casein Phosphopeptide (Recaldent ™), (Wang 2012) Tri-Calcium Phosphate ™ or Novamin ™) (Su 2011). Moreover, encouraging clinical findings have been reported, including, but not limited to the reduction of white spot enamel lesions and dentinal hypersensitivity (Kowalczyk 2006).

The topical application of "antihypersensitivity" materials is a common recommendation (least invasive of the "standard of care" recommendations) to diminish dentinal hypersensitivity and will serve to provide data for the research study. The study will evaluate which of these products result in the greatest reduction of dentinal hypersensitivity. The application of the experimental products for the reduction of dentinal hypersensitivity is for research purposes.

The methods used to test sensitivity in this study have been used in published studies (Brahmbhatt 2012, Holland 1997). The VAS scale used in this study has also been used for tooth sensitivity studies (Holland 1997, Hughes 2010). A 30% decrease in VAS score has been shown to be clinically meaningful (Ritter 2006, Raymond 2008).

This pilot study would investigate the ability of anti-caries products to reduce dentinal hypersensitivity when compared to a sensitivity-reducing dentifrice. It would be a novel contribution to the dental community if a material that is proven to reduce tooth decay is also proven to reduce dentinal hypersensitivity. The results may potentially have a tremendous impact on the dental community because it may provide dental professionals a scientifically-supported approach to improve the comfort and quality of life of periodontal patients (patients who are treated for gum disease/ bone loss around teeth) and increase the lifespan of teeth that undergo periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Tooth with exposed root surface and/or exposed dentin
* Tooth with a VAS score greater than or equal to 3
* No adjacent tooth/teeth with sensitivity (as defined as 2 or higher on the VAS)

Exclusion Criteria:

* Participation in another dental study that may alter the results of this study.
* A medical condition that could interfere with reliable pain reporting (e.g., pain disorders)
* Any chronic medical condition that requires the regular use of pain or anti-inflammatory medications
* Used a desensitizing dentifrice within the preceding four weeks
* Have received an antihypersensitivity treatment (varnish or precipitating solution) of the identified tooth within the preceding four weeks
* Undergoing active orthodontic treatment.
* Teeth with carious lesions, buccal vertical cracks in enamel, evidence of irreversible pulpitis (pain lasting more than five seconds after air stimulation)
* Pregnant/ lactating patients (Clinpro5000 has 5000ppm fluoride and there is a risk of ingesting the product)
* Patients with Milk Allergy (CPP-ACP is a dairy based product)
* Patients on Kidney Dialysis (due to the free calcium in CPP-ACP, dialysis patients should be on a diet with limited calcium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-05; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britta Magnuson, DMD, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pradeep AR, Sharma A. Comparison of clinical efficacy of a dentifrice containing calcium sodium phosphosilicate to a dentifrice containing potassium nitrate and to a placebo on dentinal hypersensitivity: a randomized clinical trial. J Periodontol. 2010 Aug;81(8):1167-73. doi: 10.1902/jop.2010.100056. PMID 20370417
- [Background] Yilmaz HG, Kurtulmus-Yilmaz S, Cengiz E. Long-term effect of diode laser irradiation compared to sodium fluoride varnish in the treatment of dentine hypersensitivity in periodontal maintenance patients: a randomized controlled clinical study. Photomed Laser Surg. 2011 Nov;29(11):721-5. doi: 10.1089/pho.2010.2974. Epub 2011 Jun 13. PMID 21668343
- [Background] West NX. Dentine hypersensitivity: preventive and therapeutic approaches to treatment. Periodontol 2000. 2008;48:31-41. doi: 10.1111/j.1600-0757.2008.00262.x. No abstract available. PMID 18715354
- [Background] Saunders RH Jr, Meyerowitz C. Dental caries in older adults. Dent Clin North Am. 2005 Apr;49(2):293-308. doi: 10.1016/j.cden.2004.10.004. PMID 15755406
- [Background] Hull PS, Worthington HV, Clerehugh V, Tsirba R, Davies RM, Clarkson JE. The reasons for tooth extractions in adults and their validation. J Dent. 1997 May-Jul;25(3-4):233-7. doi: 10.1016/s0300-5712(96)00029-2. PMID 9175351
- [Background] Brahmbhatt N, Bhavsar N, Sahayata V, Acharya A, Kshatriya P. A double blind controlled trial comparing three treatment modalities for dentin hypersensitivity. Med Oral Patol Oral Cir Bucal. 2012 May 1;17(3):e483-90. doi: 10.4317/medoral.17594. PMID 22143734
- [Background] Orsini G, Procaccini M, Manzoli L, Giuliodori F, Lorenzini A, Putignano A. A double-blind randomized-controlled trial comparing the desensitizing efficacy of a new dentifrice containing carbonate/hydroxyapatite nanocrystals and a sodium fluoride/potassium nitrate dentifrice. J Clin Periodontol. 2010 Jun;37(6):510-7. doi: 10.1111/j.1600-051X.2010.01558.x. PMID 20507374
- [Background] Jenson L, Budenz AW, Featherstone JD, Ramos-Gomez FJ, Spolsky VW, Young DA. Clinical protocols for caries management by risk assessment. J Calif Dent Assoc. 2007 Oct;35(10):714-23. PMID 18044379
- [Background] Young DA, Featherstone JD, Roth JR, Anderson M, Autio-Gold J, Christensen GJ, Fontana M, Kutsch VK, Peters MC, Simonsen RJ, Wolff MS. Caries management by risk assessment: implementation guidelines. J Calif Dent Assoc. 2007 Nov;35(11):799-805. PMID 18080486
- [Background] Featherstone JD, Zero DT. An in situ model for simultaneous assessment of inhibition of demineralization and enhancement of remineralization. J Dent Res. 1992 Apr;71 Spec No:804-10. doi: 10.1177/002203459207100S02. PMID 1592963
- [Background] Ito A, Hayashi M, Hamasaki T, Ebisu S. How regular visits and preventive programs affect onset of adult caries. J Dent Res. 2012 Jul;91(7 Suppl):52S-58S. doi: 10.1177/0022034511435701. PMID 22699669
- [Background] Wang JX, Yan Y, Wang XJ. Clinical evaluation of remineralization potential of casein phosphopeptide amorphous calcium phosphate nanocomplexes for enamel decalcification in orthodontics. Chin Med J (Engl). 2012 Nov;125(22):4018-21. PMID 23158136
- [Background] Su N, Marek CL, Ching V, Grushka M. Caries prevention for patients with dry mouth. J Can Dent Assoc. 2011;77:b85. PMID 21774875
- [Background] Kowalczyk A, Botulinski B, Jaworska M, Kierklo A, Pawinska M, Dabrowska E. Evaluation of the product based on Recaldent technology in the treatment of dentin hypersensitivity. Adv Med Sci. 2006;51 Suppl 1:40-2. PMID 17458057
- [Background] Holland GR, Narhi MN, Addy M, Gangarosa L, Orchardson R. Guidelines for the design and conduct of clinical trials on dentine hypersensitivity. J Clin Periodontol. 1997 Nov;24(11):808-13. doi: 10.1111/j.1600-051x.1997.tb01194.x. PMID 9402502
- [Background] Hughes N, Mason S, Jeffery P, Welton H, Tobin M, O'Shea C, Browne M. A comparative clinical study investigating the efficacy of a test dentifrice containing 8% strontium acetate and 1040 ppm sodium fluoride versus a marketed control dentifrice containing 8% arginine, calcium carbonate, and 1450 ppm sodium monofluorophosphate in reducing dentinal hypersensitivity. J Clin Dent. 2010;21(2):49-55. PMID 20669816
- [Background] Ritter AV, de L Dias W, Miguez P, Caplan DJ, Swift EJ Jr. Treating cervical dentin hypersensitivity with fluoride varnish: a randomized clinical study. J Am Dent Assoc. 2006 Jul;137(7):1013-20; quiz 1029. doi: 10.14219/jada.archive.2006.0324. PMID 16803829
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Teeth
Period: Overall Study
Arm/Group | Sensodyne | Crest Cavity Protection & MI Paste Plus | Clinpro 5000
Started | 13; 13 Teeth | 13; 13 Teeth | 13; 13 Teeth
Completed | 11; 11 Teeth | 13; 13 Teeth | 13; 13 Teeth
Not Completed | 2; 2 Teeth | 0; 0 Teeth | 0; 0 Teeth
Not completed — Lost to Follow-up | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Teeth
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensodyne | Crest Cavity Protection & MI Paste Plus | Clinpro 5000 | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Number analyzed (Teeth) | 13 | 13 | 13 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 13 | 37
  >=65 years | 0 | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.08 (7.99) | 45.62 (15.23) | 45.85 (13.64) | 48.85 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 7 | 24
  Male | 5 | 4 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 4 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 4 | 11
  White | 6 | 6 | 3 | 15
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 13 | 39
Baseline Dentinal Hypersensitivity [Median (Inter-Quartile Range); unit: units on a scale] — Air test: 1 sec blast of air from air-water syringe was applied
  Water test: 3 drops of ice water were applied
  Schiff Score Investigator observed participant reaction to test and scored
  0-Subject does not respond to stimulus
  1. Subject responds to stimulus, but does not request discontinuation of stimulus
  2. Subject responds to stimulus and requests discontinuation or moves from stimulus
  3. Subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus
  VAS Participant reported sensitivity on scale. 0-no pain, 10-worst pain imaginable
  units on a scale
    Air Schiff | 1 [0 to 1] | 1 [1 to 1] | 1 [1 to 2] | 1 [1 to 2]
    Air VAS | 5 [4 to 7] | 5 [4 to 8] | 5 [4 to 6] | 5 [4 to 7]
    Water Schiff | 1 [0 to 2] | 1 [0 to 2] | 1 [1 to 2] | 1 [1 to 2]
    Water VAS | 6 [4 to 7] | 6 [5 to 7] | 6 [5 to 8] | 6 [4.5 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Dentinal Hypersensitivity
Description: The primary analysis will be to compare the dentinal hypersensitivity between the 3 groups.
  Air test: A 1 second blast of air from the air-water syringe was applied to the tooth.
  Water test: Three drops of ice water were be placed on the tooth.
  Schiff Score
  Investigator observed participant reaction to test and scored on following scale:
  0-Tooth/Subject does not respond to stimulus.
  1. Tooth/Subject responds to stimulus, but does not request discontinuation of stimulus.
  2. Tooth/Subject responds to stimulus and requests discontinuation or moves from stimulus.
  3. Tooth/Subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus
  VAS (visual analog scale):
  The participant reported sensitivity on a scale of 0-10. 0 being no pain and 10 being worst pain imaginable.
Time Frame: 8 weeks after baseline
Measure: Median (Inter-Quartile Range); unit: units on a scale
Units Other Than Participants: Teeth
Arm/Group | Sensodyne | Crest Cavity Protection & MI Paste Plus | Clinpro 5000
Number analyzed (Participants) | 11 | 13 | 13
Number analyzed (Teeth) | 11 | 13 | 13
units on a scale
  Air Schiff | 1 [0 to 1] | 1 [0 to 1] | 0 [0 to 1]
  Air VAS | 3 [0.5 to 4] | 2 [1 to 3] | 2 [1 to 3]
  Water Schiff | 1 [0 to 1] | 1 [0 to 1] | 1 [0 to 1]
  Water VAS | 4 [2.5 to 5.5] | 2 [1 to 3] | 2 [1 to 5]
Statistical Analysis 1: Comparison: Sensodyne vs Crest Cavity Protection & MI Paste Plus vs Clinpro 5000; Assuming the control group may exhibit a modest improvement in dentinal hypersensitivity (~5%) whereas the two test groups should demonstrate a more significant improvement (~30%). Assuming a common standard deviation of 25%, we will have 58% power to detect a difference between the 3 groups using one way analysis of variance, with 10 subjects per group, and setting alpha to 0.05 (nQuery Advisor, Version 7.0). Up to 13 subjects per group will be recruited, to allow for a 20% dropout rate; Test type: Superiority; p = 0.72, Kruskal-Wallis — This p-value is for the Air Schiff comparison. The threshold of significance was 0.05 and no multiple comparisons were necessary
Statistical Analysis 2: Comparison: Sensodyne vs Crest Cavity Protection & MI Paste Plus vs Clinpro 5000; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .93, Kruskal-Wallis — This p-value is for the Air VAS comparison. The threshold of significance was 0.05 and no multiple comparisons were necessary
Statistical Analysis 3: Comparison: Sensodyne vs Crest Cavity Protection & MI Paste Plus vs Clinpro 5000; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .77, Kruskal-Wallis — This p-value is for the WaterSchiff comparison. The threshold of significance was 0.05 and no multiple comparisons were necessary
Statistical Analysis 4: Comparison: Sensodyne vs Crest Cavity Protection & MI Paste Plus vs Clinpro 5000; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .93, Kruskal-Wallis — This p-value is for the WaterVAS comparison. The threshold of significance was 0.05 and no multiple comparisons were necessary

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Sensodyne | Crest Cavity Protection & MI Paste Plus | Clinpro 5000
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 2/13 | 3/13 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sensodyne (N=13) | Crest Cavity Protection & MI Paste Plus (N=13) | Clinpro 5000 (N=13)
Headache (Nervous system disorders) | 0 | 0 | 1
Infection of foot (Infections and infestations) | 1 | 0 | 0 — Subject cut foot and had subsequent infection
Skin finding (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Swelling/bump on subject's back
Fracture of tooth (Injury, poisoning and procedural complications) | 0 | 1 | 0
Accidental fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 — Subject accidentally fell and bruised ribs
Migraine (Nervous system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT02136576/Prot_SAP_000.pdf